CLINICAL TRIAL: NCT06675201
Title: Neoantigen Vaccines in Combination with Immune Checkpoint Inhibitors for Maintenance Therapy Following Definitive Treatment of Locally Advanced Unresectable Esophageal Squamous Cell Carcinoma: an Open-Label, Randomized, Phase II Study
Brief Title: Neoantigen Vaccines in Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Clinical Professor, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHANT-241 Study
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC); Neoantigen-loaded Dendritic Cell Vaccine; Immune Checkpoint Inhibitors (ICIs)
Keywords: Esophageal Squamous Cell Carcinoma (ESCC); neoantigen tumor vaccine; immunotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NeoDC-Vac + ICIs (Experimental): Experimental Group: NeoDC-Vac combined with ICIs NeoDC-Vac: Administered via subcutaneous injections at multiple sites, including bilateral axillary and bilateral inguinal regions. The initial phase consists of 5 injections during the first cycle, given at weeks 1, 2, 4, 6, and 8. Thereafter, the vaccine is administered once every 4 weeks, continuing for 1 year, or until disease progression, intolerable adverse events, or death from any cause.
  ICIs: Administered intravenously once a month, with a maintenance duration of 1 year, or until disease progression, intolerable adverse events, or death from any cause.
  Interventions: Biological: neoantigen-loaded dendritic cell vaccine (NeoDC-Vac)
- ICIs (Active Comparator): ICIs: Administered intravenously once a month, with a maintenance duration of 1 year, or until disease progression, intolerable adverse events, or death from any cause.
  Interventions: Biological: neoantigen-loaded dendritic cell vaccine (NeoDC-Vac)

INTERVENTIONS:
Biological: neoantigen-loaded dendritic cell vaccine (NeoDC-Vac) — Experimental Group: Neoantigen Vaccine Combined with Immune Checkpoint Inhibitors (ICIs) Neoantigen Vaccine: Administered via subcutaneous injections at multiple sites, including bilateral axillary and bilateral inguinal regions. The initial phase consists of 5 injections during the first cycle, given at weeks 1, 2, 4, 6, and 8. Thereafter, the vaccine is administered once every 4 weeks, continuing for 1 year, or until disease progression, intolerable adverse events, or death from any cause.
  ICIs: Administered intravenously once a month, with a maintenance duration of 1 year, or until disease progression, intolerable adverse events, or death from any cause.
  Control Group: ICIs ICIs: Administered intravenously once a month, with a maintenance duration of 1 year, or until disease progression, intolerable adverse events, or death from any cause.

SUMMARY:
The aim of this clinical trial is to evaluate the efficacy and safety of consolidation therapy with a neoantigen-loaded dendritic cell vaccine (NeoDC-Vac) following radical chemoradiotherapy or chemoradiation-immunotherapy in patients with locally advanced, unresectable ESCC. The primary endpoint of the study is the OS rate. Secondary endpoints include OS, PFS, adverse events, CR rate, and quality of life (QoL) of patients. Exploratory endpoints involve the assessment of biomarkers such as TMB, PD-L1, and ctDNA.

The key questions this study aims to answer are:

-Can the combination of (ICIs and NeoDC-Vac as maintenance therapy improve OS and QoL in patients with locally advanced, unresectable ESCC following radical treatment? Can this novel approach provide an effective treatment option for these patients?

Participant Procedures:

1. Endoscopic examination at West China Hospital. Baseline fresh tumor tissue collection for NGS in neoantigen vaccine group.
2. Screening assessments, informed consent, and random assignment to experimental or control group.

   Experimental Group**: Neoantigen-loaded vaccine + standard ICIs as maintenance therapy.

   Control Group**: Standard ICIs as maintenance. One cycle per month for one year.
3. Tumor tissue NGS, ctDNA analysis, TIME evaluation, T cell response profiling. All costs covered by research funding.
4. After completing the full treatment regimen, participants will be monitored with regular follow-up visits by healthcare professionals to assess ongoing health outcomes and safety.

DETAILED DESCRIPTION:
The objective of this clinical trial is to evaluate the efficacy and safety of neoantigen-loaded dendritic cell (DC) vaccines as consolidation therapy following definitive chemoradiotherapy or radiotherapy with immunotherapy in patients with locally advanced unresectable esophageal squamous cell carcinoma (ESCC). The primary endpoint is the 2-year overall survival (OS) rate. Secondary endpoints include OS, progression-free survival (PFS), adverse events, complete response (CR) rate, and patient quality of life. Exploratory endpoints focus on biomarker analysis, including tumor mutational burden (TMB), PD-L1 expression, and circulating tumor DNA (ctDNA).

The key questions this study aims to answer are whether maintenance therapy with immune checkpoint inhibitors (ICIs) combined with neoantigen vaccines can improve overall survival and quality of life in patients with locally advanced, unresectable ESCC following definitive treatment, ultimately providing a new therapeutic strategy for these patients.

**Participants in the study will:**

1. **Diagnostic Endoscopy at West China Hospital:** Participants must undergo endoscopic examination at West China Hospital to confirm diagnosis. For patients in the neoantigen vaccine group, baseline fresh tissue samples will be obtained for next-generation sequencing (NGS) to screen for neoantigen peptides, which will be used to prepare individualized neoantigen vaccines.
2. **Enrollment and Consent:** Participants will complete relevant examinations to determine eligibility. Upon confirmation of eligibility, they will provide informed consent and undergo randomization.

   **Treatment Regimen:**
   * **Experimental Group:** Neoantigen tumor vaccine in combination with standard immune checkpoint inhibitors (ICIs) as maintenance therapy following definitive treatment.
   * **Control Group:** Standard ICIs alone as maintenance therapy.

   The treatment cycle will consist of monthly administrations for a total duration of one year.
3. **Assessments During Treatment:** Key assessments during treatment will include NGS sequencing of tumor tissue, ctDNA analysis from blood samples, evaluation of the tumor immune microenvironment (TIME), and T-cell response analysis. All of these assessments are essential for receiving the study treatment, and the associated costs will be covered by the research grant, ensuring that participants incur no additional financial burden.

ELIGIBILITY:
Inclusion Criteria:

A. Age 18-80 years

B. Locally advanced unresectable ESCC patients after radical treatment (radical chemoradiotherapy or chemoradiation); including:

* Cervical esophageal segment, T4, supraclavicular lymph node metastasis, or inability/refusal to undergo surgery due to personal reasons (refer to hospital below); ② Failure of neoadjuvant or conversion therapy; ③ Postoperative local recurrence, unresectable (target lesion present). C. No evidence of tumor recurrence or metastasis 2-3 weeks after radical treatment D. Ability to provide fresh tumor tissue samples (baseline) E. Normal major organ function F. Performance status (PS) score ≤ 1 G. Patients of childbearing potential must use contraception H. Voluntary participation with signed informed consent

Exclusion Criteria:

A. History of fistula caused by primary tumor invasion B. High risk of gastrointestinal bleeding, esophageal fistula, or esophageal perforation C. Poor nutritional status D. Immune-related adverse events during prior radical treatment, such as Grade ≥3 pneumonitis, myocarditis, etc.

E. Signs and symptoms of interstitial diseases F. Presence of any severe and/or uncontrolled medical conditions G. Presence of concurrent malignancies H. Presence of other autoimmune diseases, or prolonged use of immunosuppressants or steroids I. Difficulty in patient communication or inability to comply with long-term follow-up J. Other conditions deemed unsuitable by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 165 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
2-year OS rate | 24months
  Overall Survival (OS) is defined as the time from randomization (following radical treatment) to death from any caus

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 12months
  The progression-free survival (PFS) is defined as the time from random assignment to the occurrence of the first event, which could be local failure, metastatic recurrence, disease progression, or death from any cause
Treatment-related adverse effects (TRAEs) | 12months
  This study will collected any adverse medical events that occurred during the study drug treatment, and the treatment-related adverse events as assessed by CTCAE v5.0.

OTHER OUTCOMES:
Biomarker analysis of tumor mutational burden (TMB) | 12months
  Whole exome sequencing (WES) will be performed on tumor tissue samples collected prior to vaccine immunization to analyze the relationship between tumor mutational burden (TMB) and the efficacy of the vaccine therapy.
Biomarker analysis of tumor circulating tumor DNA (ctDNA) | 12months
  The recurrence and metastasis of the tumor will be monitored through circulating tumor DNA (ctDNA) at four specific time points: at baseline, two weeks after the first cycle of vaccine immunization (i.e., 2.5 months post-treatment), during the vaccine boost phase (6 months post-treatment), and at the time of tumor progression.

CONTACTS AND LOCATIONS:
Overall Officials: zhenyu ding, MD, Principal Investigator — West China Hospital of Sichuan University, ChengDu, China
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Please Select, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Zheng Y, Shi H, Yang W, Xu H, Li Y, Ding Z. Personalized neoantigen DC vaccine combined with camrelizumab following definitive therapy in locally advanced unresectable esophageal squamous cell carcinoma (CHANT-241): protocol for a randomized controlled trial. Front Immunol. 2026 Jan 12;16:1658670. doi: 10.3389/fimmu.2025.1658670. eCollection 2025. PMID 41601631